CLINICAL TRIAL: NCT02294110
Title: Phase IV Study of Diabetes Mellitus for Spinal Anesthesia Failure
Brief Title: Effect of Diabetes Mellitus on Success of Spinal Anesthesia
Status: Completed | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, İBRAHİM ÖZTÜRK, phase IV study of diabetes mellitus for spinal anesthesia failure, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: DMSAFAILURE
Record Dates: First submitted 2014-10-12; First posted 2014-11-19 (Estimated); Last update posted 2015-08-05 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes Mellitus
Keywords: failure; spinal anesthesia
MeSH Terms: conditions — Diabetes Mellitus | interventions — Anesthesia, Spinal

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- diabetes mellitus: spinal anesthesia
  Interventions: Other: spinal anesthesia

INTERVENTIONS:
Other: spinal anesthesia — non diabetes mellitus

SUMMARY:
Some of the authors says that diabetes mellitus is a risk factor for spinal anesthesia failure. However, that opinion was not determined in a trial. Thus the investigators aimed to investigate the effect of diabetes mellitus on spinal anesthesia.

DETAILED DESCRIPTION:
The investigators will include all of the patients who will undergo surgery with spinal anesthesia. The investigators will observe the patients with or without diabetes mellitus. And the investigators will examine the effect of diabetes mellitus on failure of spinal anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* surgery with spinal anesthesia

Exclusion Criteria:

* heart failure
* coronary artery disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients who undergoes surgery with spinal anesthesia
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2014-11; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
sensorial loss with pin prick test | intraoperative 5 th minute

CONTACTS AND LOCATIONS:
Overall Officials: dilek yazıcıoğlu, M.D., Study Chair — M.D.

REFERENCES:
- [Background] Hoppe J, Popham P. Complete failure of spinal anaesthesia in obstetrics. Int J Obstet Anesth. 2007 Jul;16(3):250-5. doi: 10.1016/j.ijoa.2006.12.005. Epub 2007 May 16. PMID 17509868